CLINICAL TRIAL: NCT04565652
Title: Clinical Evaluation of the LOIS Smartband in Patients Undergoing Elective ICD Implantation With Defibrillation (DFT) Threshold Testing.
Brief Title: ICD Shock Detection by a Wearable
Acronym: LOISICD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lois Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 264962
Record Dates: First submitted 2020-09-10; First posted 2020-09-25 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Arrest; Heart Arrest; Cardiopulmonary Arrest
Keywords: ICD; Defibrillator
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: A single group of patients will wear the LOIS ICD smartband during elective ICD defibrillation
Masking Description: Each patient will knowingly wear the ICD Smartband
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICD Defibrillation (Experimental): Detection of ICD shock during elective ICD implant using the investigational device
  Interventions: Device: Device Wearers

INTERVENTIONS:
Device: Device Wearers — The intervention arm will wear the LOIS ICD Smartband during routine ICD defibrillation following elective ICD implant.

SUMMARY:
Trial to assess the ability of a wearable to detect defibrillation from an implantable ICD

DETAILED DESCRIPTION:
Non-invasive, pain-free clinical evaluation of a wearable/proximity sensor designed to detect a high voltage therapeutic shock received by a patient from their Implantable Cardioverter Defibrillator (ICD) during defibrillation threshold testing (DFT), which is a routine part of the clinical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding procedure and making informed consent
* Listed for elective ICD Implant
* Having routine DFT as part of elective ICD implantation

Exclusion Criteria:

* Not indicated for ICD implant
* Incapable of making informed consent
* Pregnant
* Not on stabilised anti-coagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of investigational device at detecting ICD shocks | 1 year
  The number of successful detection of ICD shocks using the novel ICD Smartband versus missed events

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom